CLINICAL TRIAL: NCT03799003
Title: A Phase 1b Study of ASP1951, a GITR Agonistic Antibody, as a Single Agent and in Combination With Pembrolizumab in Subjects With Advanced Solid Tumors
Brief Title: A Study of ASP1951 in Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated for lack of efficacy.
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1951-CL-0101; 2019-002287-27 (EudraCT Number); KEYNOTE-B02 (Other: Merck); MK-3475-B02 (Other: Merck)
Record Dates: First submitted 2019-01-02; First posted 2019-01-10 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Advanced Solid Tumors
Keywords: ASP1951; cervical cancer; Oncology; squamous cell carcinoma of the head and neck (SCCHN); metastatic castration-resistant prostate cancer (mCRPC); melanoma; Tumors; pembrolizumab; colorectal cancer; Advanced (unresectable) or metastatic solid tumor malignancies; Advanced solid tumors
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasms; Squamous Cell Carcinoma of Head and Neck; Melanoma; Colorectal Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- ASP1951 0.07 mg Monotherapy (Experimental): Participants have received ASP1951 0.07 mg intravenously on day 1 of every 3-week cycle.
  Interventions: Drug: ASP1951
- ASP1951 0.7 mg Monotherapy (Experimental): Participants have received ASP1951 0.7 mg intravenously on day 1 of every 3-week cycle.
  Interventions: Drug: ASP1951
- ASP1951 5 mg Monotherapy (Experimental): Participants have received ASP1951 5 mg intravenously on day 1 of every 3-week cycle.
  Interventions: Drug: ASP1951
- ASP1951 20 mg Monotherapy (Experimental): Participants have received ASP1951 20 mg intravenously on day 1 of every 3-week cycle.
  Interventions: Drug: ASP1951
- ASP1951 70 mg Monotherapy (Experimental): Participants have received ASP1951 70 mg intravenously on day 1 of every 3-week cycle.
  Interventions: Drug: ASP1951
- ASP1951 200 mg Monotherapy (Experimental): Participants have received ASP1951 200 mg intravenously on day 1 of every 3-week cycle.
  Interventions: Drug: ASP1951
- ASP1951 700 mg Monotherapy (Experimental): Participants have received ASP1951 700 mg intravenously on day 1 of every 3-week cycle.
  Interventions: Drug: ASP1951
- ASP1951 1400 mg Monotherapy (Experimental): Participants have received ASP1951 1400 mg intravenously on day 1 of every 3-week cycle.
  Interventions: Drug: ASP1951
- ASP1951 20 mg + pembrolizumab 200 mg Combination Therapy (Experimental): Participants have received ASP1951 20 mg intravenously on day 1 of every 3-week cycle in combination with pembrolizumab 200 mg administered on day 1 of every 3-week cycle, at least 30 minutes after the end of infusion of ASP1951.
  Interventions: Drug: ASP1951; Drug: pembrolizumab
- ASP1951 700 mg + pembrolizumab 200 mg Combination Therapy (Experimental): Participants have received ASP1951 700 mg intravenously on day 1 of every 3-week cycle in combination with pembrolizumab 200 mg administered on day 1 of every 3-week cycle, at least 30 minutes after the end of infusion of ASP1951.
  Interventions: Drug: ASP1951; Drug: pembrolizumab
- ASP1951 1400 mg + pembrolizumab 200 mg Combination Therapy (Experimental): Participants have received ASP1951 1400 mg intravenously on day 1 of every 3-week cycle in combination with pembrolizumab 200 mg administered on day 1 of every 3-week cycle, at least 30 minutes after the end of infusion of ASP1951.
  Interventions: Drug: ASP1951; Drug: pembrolizumab

INTERVENTIONS:
Drug: ASP1951 — Intravenously (IV)
Drug: pembrolizumab — Intravenously (IV)
  Other Names: KEYTRUDA®
  Arms: ASP1951 1400 mg + pembrolizumab 200 mg Combination Therapy; ASP1951 20 mg + pembrolizumab 200 mg Combination Therapy; ASP1951 700 mg + pembrolizumab 200 mg Combination Therapy

SUMMARY:
The primary purpose of this study is to evaluate the tolerability and safety profile of ASP1951 when administered as a single agent and in combination with pembrolizumab in participants with locally advanced (unresectable) or metastatic solid tumors; characterize the pharmacokinetic profile of ASP1951 when administered as a single agent and in combination with pembrolizumab; and determine the recommended phase 2 dose (RP2D) of ASP1951 and/or maximum tolerated dose (MTD) when administered as a single agent and in combination with pembrolizumab. This study will also evaluate the anti-tumor effect of ASP1951 when administered as a single agent and in combination with pembrolizumab.

DETAILED DESCRIPTION:
This is a dose-escalation and expansion study of ASP1951. The study consists of 3 periods for monotherapy and combination therapy: screening, treatment and follow up, followed by an optional Re-treatment period for participants that qualify.

The monotherapy escalation cohorts will evaluate escalating dose levels of ASP1951 in participants with locally advanced (unresectable) or metastatic solid tumor malignancies including but not limited to squamous cell carcinoma of the head and neck (SCCHN), colorectal cancer, metastatic castration-resistant prostate cancer (mCRPC) and cervical cancer.

The combination escalation cohorts will evaluate escalating dose levels of ASP1951 in combination with a fixed dose of pembrolizumab.

For dose expansion, the tumor-specific cohorts will include participants with squamous cell carcinoma of the head and neck (SCCHN), non-small cell lung cancer (NSCLC) (all PD-L1 status), NSCLC PDL1 high, and cervical cancer, as well as participants with any tumor types that respond to study drug treatment during dose escalation.

Participants may reinitiate study drug treatment in the optional Re-treatment period after confirmation that the participant meets all the re-treatment eligibility criteria.

After discontinuation of study drug, all participants will complete an end-of-treatment visit, along with 30-day and 90 day safety follow-up visits from the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Subject has locally-advanced (unresectable) or metastatic solid tumor malignancy (no limit to the number of prior treatment regimens) that is confirmed by available pathology records or current biopsy as well as the following:

  * Subject in the escalation cohort has received all standard therapies (unless the therapy is contraindicated or intolerable) felt to provide clinical benefit the subject's specific tumor type. OR
  * Subject in an expansion cohort has received at least 1 standard therapy for the subject's specific tumor type.

[Taiwan only]: Subject has locally-advanced (unresectable) or metastatic solid tumor malignancy (no limit to the number of prior treatment regimens) that is confirmed by available pathology records or current biopsy and has received all standard therapies (unless the therapy is contraindicated or intolerable) felt to provide clinical benefit in the opinion of the treating investigator for his/her specific tumor type. Note: Subjects in the combination expansion cohort with tumor types that pembrolizumab is not approved for can only enroll if their standard treatment is ineffective, unsuitable per investigator's judgment or if the subject is unwilling to receive the standard therapy.

* Subject has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Subject's last dose of prior antineoplastic therapy, including any immunotherapy, was 21 days or 5-half-lives, whichever is shorter, prior to initiation of study drug administration. A subject with epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) mutation-positive NSCLC is allowed to remain on EGFR tyrosine kinase inhibitor (TKI) or ALK inhibitor therapy until 4 days prior to the start of study drug administration.
* Subject has completed any radiotherapy (including stereotactic radiosurgery) at least 2 weeks prior to study drug administration. Subjects must have recovered from all radiation related toxicities, not require corticosteroids and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to noncentral nervous system [CNS] disease.
* Subject's AEs (excluding alopecia) from prior therapy have improved to grade 1 or baseline within 2 weeks prior to start of study treatment.
* Subject with metastatic castration-resistant prostate cancer (mCRPC) (positive bone scan and/or soft tissue disease documented by computed tomography [CT]/magnetic resonance imaging [MRI]) meets both of the following:

  * Subject has serum testosterone ≤ 50 ng/dL at Screening.
  * Subject has had a bilateral orchiectomy or plans to continue androgen deprivation therapy (ADT) for the duration of study treatment.
* Subject has adequate organ function prior to start of study treatment. If a subject has received a recent blood transfusion, the laboratory tests must be obtained ≥ 4 weeks after any blood transfusion. Subjects can be on stable dose of erythropoietin (≥ approximately 3 months).
* A female subject is eligible to participate if she is not pregnant and at least 1 of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP); OR
  * WOCBP who agrees to follow the contraceptive guidance throughout the treatment period and for at least 6 months after the final study drug administration.
* Female subject must agree not to breastfeed starting at Screening and throughout the study treatment, and for 6 months after the final study drug administration.
* Female subject must not donate ova starting at Screening and throughout the study treatment, and for 6 months after the final study drug administration.
* A male subject with female partner(s) of childbearing potential must agree to use contraception during the treatment period and for at least 6 months after the final study drug administration.
* A male subject must not donate sperm during the treatment period and for at least 6 months after the final study drug administration.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner is breastfeeding throughout the study period and for 6 months after the final study drug administration.
* Subject agrees not to participate in another interventional study while receiving study drug (Subjects who are currently in the follow-up period of an interventional clinical trial are allowed).

Additional Inclusion Criteria for Subjects in the Expansion Cohorts:

* Subject has at least 1 measureable lesion per RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions. Subjects with mC RPC who do not have measurable lesions must have at least 1 of the following:

  * Progression with 2 or more new bone lesions; or
  * Prostate-specific antigen (PSA) progression (defined as a minimum of 3 rising PSA levels with an interval of ≥ 1 week between each determination) within 6 weeks prior to study drug administration and a PSA value at the screening visit ≥ 2 ng/mL.
* Subject consents to provide available tumor specimen in a tissue block or unstained serial slides obtained within 56 days prior to first dose of study treatment. Note: This does not apply to subjects with mCRPC who do not have measurable disease.
* Subject is an appropriate candidate for tumor biopsy and consents to undergoing a tumor biopsy (core needle biopsy or excision) during the treatment period as indicated in the Schedule of Assessments. Note: This does not apply to subjects with mCRPC who do not have measurable disease.
* Subject meets one of the following:

  * Subject has the tumor type for which a confirmed response was observed in a monotherapy or combination therapy cohort; or
  * Subject has SCCHN and a combination therapy expansion cohort is opened due to achieving the predicted efficacious exposure or
  * High dose RP2D combination therapy expansion cohorts are opened and subject has NSCLC (all PD-L1 status), NSCLC PD-L1 high*, SCCHN, or cervical cancer; or
  * Low dose RP2D combination therapy expansion cohorts are opened and subject has NSCLC (all PD-L1 status), SCCHN and cervical cancer.

    * NSCLC with PD-L1 high expressing tumor (tumor proportion score ≥ 50%) as determined by 22C3 PD-L1 immunohistochemistry assay at a local/central laboratory during the screening period. Note: Local 22C3 PD-L1 IHC assay results available within 60 days prior study drug administration may be used for evaluating this entry criterion.

Additional Inclusion Criteria for Re-treatment:

* Subject stopped initial treatment with ASP1951 or ASP1951 in combination with pembrolizumab after attaining a confirmed CR, PR or SD.
* Subject experienced an investigator-determined iCPD after stopping their initial treatment with ASP1951 or ASP1951 in combination with pembrolizumab.
* Subject did not receive any prohibited anti-cancer treatment since the last dose of ASP1951 or ASP1951 in combination with pembrolizumab.
* Subject did not experience a toxicity that met treatment discontinuation criteria during the initial treatment with ASP1951 or ASP1951 in combination with pembrolizumab or pembrolizumab alone.

Exclusion Criteria:

* Subject weighs < 45 kg.
* Subject has received investigational therapy (other than an investigational EGFR TKI in a subject with EGFR activating mutations or ALK inhibitor in a subject with an ALK mutation) within 21 days or 5-half-lives, whichever is shorter, prior to start of study drug.
* Subject requires or has received systemic steroid therapy or any other immunosuppressive therapy within 14 days prior to study drug administration. Subjects using a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 30 mg per day of hydrocortisone, 2 mg per day of dexamethasone, or up to 10 mg per day of prednisone) are allowed.
* Subject has symptomatic CNS metastases or subject has evidence of unstable CNS metastases even if asymptomatic (e.g., progression on scans). Subjects with previously treated CNS metastases are eligible, if they are clinically stable and have no evidence of CNS progression by imaging for at least 4 weeks prior to start of study treatment and are not requiring immunosuppressive doses of systemic steroids (> 30 mg per day of hydrocortisone, > 2 mg per day of dexamethasone, or > 10 mg per day of prednisone or equivalent) for longer than 2 weeks.
* Subject has leptomeningeal disease as a manifestation of the current malignancy.
* Subject has an active autoimmune disease that has required systemic treatment in the past 2 years. Subjects with type 1 diabetes mellitus, endocrinopathies stably maintained on appropriate replacement therapy, and skin disorders (e.g., vitiligo, psoriasis or alopecia) not requiring systemic treatment are allowed.
* Subject was discontinued from prior immunomodulatory therapy due to a grade ≥ 3 toxicity that was mechanistically related (e.g., immune related) to the agent.
* Subject has known history of serious hypersensitivity reaction (≥ grade 3) to a known ingredient of ASP1951 or pembrolizumab or severe hypersensitivity reaction to treatment with another monoclonal antibody.
* Subject with positive Hepatitis B virus (HBV) antibodies and surface antigen (indicating acute HBV or chronic HBV) or Hepatitis C ([HCV]; ribonucleic acid [RNA] detected by qualitative or quantitative assay). Hepatitis C RNA testing is not required in subjects with negative Hepatitis C antibody testing. HBV antibodies are not required in subjects with negative HBV surface antigen.
* Subject has received a live vaccine against infectious diseases within 4 weeks prior to initiation of study treatment.
* Subject has a history of drug-induced pneumonitis (interstitial lung disease), a history of (non-infectious) pneumonitis that required steroids, radiation pneumonitis or currently has pneumonitis.
* Subject has an infection requiring systemic therapy within 2 weeks prior to study drug administration.
* Subject has received a prior allogeneic bone marrow or solid organ transplant.
* Subject is expected to require another form of antineoplastic therapy while on study treatment.
* Subject has had a myocardial infarction or unstable angina within 6 months prior to the start of study treatment or currently has an uncontrolled illness including, but not limited to symptomatic congestive heart failure, clinically significant cardiac disease, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subject has received prior treatment with an anti-glucocorticoid-induced tumor necrosis factor receptor (GITR) antibody.
* Subject has had a major surgical procedure and has not completely recovered within 28 days prior to the start of study treatment.
* Subject has any condition which makes the subject unsuitable for study participation.
* Subject has a known history of human immunodeficiency virus (HIV) infection. No HIV testing is required unless mandated by local health authority.
* Subject has known history of coronavirus disease 2019 (COVID-19) positive polymerase chain reaction (PCR) test within 4 weeks prior to start of study treatment.

Additional Exclusion Criterion for Subjects in Expansion Cohorts:

* Subject has a prior malignancy, other than the current malignancy for which the subject is seeking treatment, active (i.e., requiring treatment of intervention) within the previous 2 years except for locally curable malignancies that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix or breast.

Additional Exclusion Criteria for Re-treatment:

* Subjects who have completed 45 weeks in monotherapy or 57 weeks in combination therapy follow-up with disease control are not eligible for re-treatment.
* Subject currently has an ongoing AE related to ASP1951 or ASP1951 in combination with pembrolizumab that meets the criteria for treatment interruption or discontinuation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed by Dose Limiting Toxicity (DLT) | Up to 5 years
  A DLT is defined as any of the prespecified Adverse Events (AEs) (graded using National Cancer Institute Common Terminology Criteria for Adverse Events [NCI-CTCAE] version 4.03) that the investigator (or sponsor) cannot clearly attribute to a cause other than study drug.
Safety and tolerability assessed by adverse events (AEs) | Up to 5 years
  Initial and retreatment. An AE is any untoward medical occurrence in a participant administered a study drug, and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product whether or not considered related to the medicinal product. AEs will be coded using the medical dictionary for regulatory activities (MedDRA) and graded using NCI-CTCAE 4.03.
Safety and tolerability assessed by immune-related AEs (irAEs) | Up to 5 years
  Initial and retreatment. Most frequent immune-related AEs include rash, oral mucositis, dry mouth, colitis/diarrhea, hepatitis, pneumonitis, and endocrinopathies (hypophysitis, hypothyroidism, hyperthyroidism, adrenal insufficiency and Type 1 diabetes mellitus). In the event a participant is diagnosed with an irAE, then it should be reported as an AE.
Safety and tolerability assessed by infusion-related reactions (IRRs) | Up to 5 years
  Initial and retreatment. IRRs are considered AEs of special interest. In the event a participant is diagnosed with an IRR, then it should be reported as an AE.
Safety and tolerability assessed by serious adverse events (SAEs) | Up to 5 years
  Initial and retreatment. An AE is considered "serious" if it results in any of the following outcomes: results in death; is life-threatening; results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions; results in congenital anomaly or birth defect; requires inpatient hospitalization (except for planned procedures as allowed per study) or leads to prolongation of hospitalization (except if prolongation of planned hospitalization is not caused by an AE). Hospitalization for treatment/observation/examination caused by AE is to be considered as serious; and other medically important events.
Number of participants with laboratory value abnormalities and/or adverse events related to treatment | Up to 5 years
  Initial and retreatment. Number of participants with potentially clinically significant laboratory values.
Safety and tolerability assessed by 12- lead electrocardiogram (ECG) | Up to 5 years
  Initial and retreatment. ECGs should be obtained after the participant has rested in supine position (or semi-recumbent, if supine is not tolerated) for 10 minutes. Any clinically significant adverse changes on the ECG will be reported as AEs.
Number of participants with vital signs abnormalities and/or adverse events related to treatment | Up to 5 years
  Initial and retreatment. Number of participants with potentially clinically significant vital sign values.
Number of participants with Physical Exam abnormalities and/or adverse events related to treatment | Up to 5 years
  Initial and retreatment. Number of participants with potentially clinically significant physical exam values.
Safety and tolerability assessed by ECOG performance status | Up to 5 years
  Initial and retreatment. The Eastern Cooperative Oncology Group (ECOG) scale will be used to assess performance status. Grades range from 0 (fully active) to 4 (completely disabled). Negative change scores indicate an improvement. Positive scores indicate a decline in performance.
Pharmacokinetics (PK) of ASP1951 in serum: AUClast | Up to 10 weeks
  Initial monotherapy escalation treatment only. Area under the concentration time curve from the time of dosing to the last measurable concentration (AUClast) will be recorded from the pharmacokinetic (PK) serum samples collected.
Pharmacokinetics (PK) of ASP1951 in serum: AUCinf | Up to 10 weeks
  Initial monotherapy escalation treatment only. Area under the concentration time curve from the time of dosing extrapolated to time infinity (AUCinf) will be recorded from the pharmacokinetic (PK) serum samples collected.
Pharmacokinetics (PK) of ASP1951 in serum: AUCinf%extrap | Up to 10 weeks
  Initial monotherapy escalation treatment only. Percentage of AUCinf due to extrapolation from time of the last measurable concentration to time infinity (AUCinf %extrap) will be recorded from the pharmacokinetic (PK) serum samples collected.
Pharmacokinetics (PK) of ASP1951 in serum: AUCtau | Up to 10 weeks
  Initial monotherapy escalation treatment only. Area under the concentration time curve from the time of dosing to the start of next dosing interval (AUCtau) will be recorded from the pharmacokinetic (PK) serum samples collected.
Pharmacokinetics (PK) of ASP1951 in serum: Cmax | Up to 10 weeks
  Initial monotherapy escalation treatment only. Maximum concentration (Cmax) will be recorded from the pharmacokinetic (PK) serum samples collected.
Pharmacokinetics (PK) of ASP1951 in serum: Ctrough | Up to 48 weeks
  Initial monotherapy escalation and retreatment. Concentration immediately prior to dosing at multiple dosing (Ctrough) will be recorded from the pharmacokinetic (PK) serum samples collected.
Pharmacokinetics (PK) of ASP1951 in serum: tmax | Up to 10 weeks
  Initial monotherapy escalation treatment only. Time of the maximum concentration (tmax) will be recorded from the pharmacokinetic (PK) serum samples collected.
Pharmacokinetics (PK) of ASP1951 in serum: t 1/2 | Up to 10 weeks
  Initial monotherapy escalation treatment only. Terminal elimination half-life (t1/2) will be recorded from the pharmacokinetic (PK) serum samples collected.
Pharmacokinetics (PK) of ASP1951 in serum: tlast | Up to 10 weeks
  Initial monotherapy escalation treatment only. Time of last measurable concentration (tlast) will be recorded from the pharmacokinetic (PK) serum samples collected.
Pharmacokinetics (PK) of ASP1951 in serum: CL | Up to 10 weeks
  Initial monotherapy escalation treatment only. Total clearance after intravenous dosing (CL) will be recorded from the pharmacokinetic (PK) serum samples collected.
Pharmacokinetics (PK) of ASP1951 in serum: Vz | Up to 10 weeks
  Initial monotherapy escalation treatment only. Volume of distribution after intravenous dosing during the terminal elimination phase (Vz) will be recorded from the pharmacokinetic (PK) serum samples collected.
Pharmacokinetics (PK) of ASP1951 in serum: Vss | Up to 10 weeks
  Initial monotherapy escalation treatment only. Volume of distribution at steady state after intravenous dosing (Vss) will be recorded from the pharmacokinetic (PK) serum samples collected.
Pharmacokinetics (PK) of ASP1951 in combination with pembrolizumab in serum: AUClast | Up to 10 weeks
  Initial combination escalation treatment only. Area under the concentration time curve from the time of dosing to the last measurable concentration (AUClast) will be recorded from the pharmacokinetic (PK) serum samples collected.
Pharmacokinetics (PK) of ASP1951 in combination with pembrolizumab in serum: AUCinf | Up to 10 weeks
  Initial combination escalation treatment only. Area under the concentration time curve from the time of dosing extrapolated to time infinity (AUCinf) will be recorded from the pharmacokinetic (PK) serum samples collected.
Pharmacokinetics (PK) of ASP1951 in combination with pembrolizumab in serum: AUCinf%extrap | Up to 10 weeks
  Initial combination escalation treatment only. Percentage of AUCinf due to extrapolation from time of the last measurable concentration to time infinity (AUCinf %extrap) will be recorded from the pharmacokinetic (PK) serum samples collected.
Pharmacokinetics (PK) of ASP1951 in combination with pembrolizumab in serum: AUCtau | Up to 10 weeks
  Initial combination escalation treatment only. Area under the concentration time curve from the time of dosing to the start of next dosing interval (AUCtau) will be recorded from the pharmacokinetic (PK) serum samples collected.
Pharmacokinetics (PK) of ASP1951 in combination with pembrolizumab in serum: Cmax | Up to 10 weeks
  Initial combination escalation treatment only. Maximum concentration (Cmax) will be recorded from the pharmacokinetic (PK) serum samples collected.
Pharmacokinetics (PK) of ASP1951 in combination with pembrolizumab in serum: Ctrough | Up to 48 weeks
  Initial combination escalation and retreatment. Concentration immediately prior to dosing at multiple dosing (Ctrough) will be recorded from the pharmacokinetic (PK) serum samples collected.
Pharmacokinetics (PK) of ASP1951 in combination with pembrolizumab in serum: tmax | Up to 10 weeks
  Initial combination escalation treatment only. Time of the maximum concentration (tmax) will be recorded from the pharmacokinetic (PK) serum samples collected.
Pharmacokinetics (PK) of ASP1951 in combination with pembrolizumab in serum: t 1/2 | Up to 10 weeks
  Initial combination escalation treatment only. Terminal elimination half-life (t1/2) will be recorded from the pharmacokinetic (PK) serum samples collected.
Pharmacokinetics (PK) of ASP1951 in combination with pembrolizumab in serum: tlast | Up to 10 weeks
  Initial combination escalation treatment only. Time of last measurable concentration (tlast) will be recorded from the pharmacokinetic (PK) serum samples collected.
Pharmacokinetics (PK) of ASP1951 in combination with pembrolizumab in serum: CL | Up to 10 weeks
  Initial combination escalation treatment only. Total clearance after intravenous dosing (CL) will be recorded from the pharmacokinetic (PK) serum samples collected.
Pharmacokinetics (PK) of ASP1951 in combination with pembrolizumab in serum: Vz | Up to 10 weeks
  Initial combination escalation treatment only. Volume of distribution after intravenous dosing during the terminal elimination phase (Vz) will be recorded from the pharmacokinetic (PK) serum samples collected.
Pharmacokinetics (PK) of ASP1951 in combination with pembrolizumab in serum: Vss | Up to 10 weeks
  Initial combination escalation treatment only. Volume of distribution at steady state after intravenous dosing (Vss) will be recorded from the pharmacokinetic (PK) serum samples collected.
Recommended Phase 2 Dose (RP2D) of ASP1951 | Up to 5 years
  RP2D of ASP1951 as a single agent is determined using available data on safety, pharmacokinetics, pharmacodynamics and efficacy of ASP1951.
RP2D of ASP1951 in combination with pembrolizumab | Up to 5 years
  RP2D of ASP1951 in combination with pembrolizumab is determined using available data on safety, pharmacokinetics, pharmacodynamics and efficacy of ASP1951.
Maximum Tolerated Dose (MTD) of ASP1951 | Up to 5 years
  MTD is defined as the dose level at which the posterior mean of DLT rate estimated using Bayesian CRM is closest but does not exceed the target DLT rate of 33%, based on the profile of DLTs collected.
MTD of ASP1951 in combination with pembrolizumab | Up to 5 years
  MTD is defined as the dose level at which the posterior mean of DLT rate estimated using Bayesian CRM is closest but does not exceed the target DLT rate of 33%, based on the profile of DLTs collected.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per Response Evaluation Criteria In Solid Tumors (RECIST) V1.1 and modified RECIST 1.1 for immune-based therapeutics (iRECIST) | Up to 5 years
  Initial and retreatment. ORR is defined as the proportion of participants for each dose level whose best overall response is rated as confirmed complete response (CR) or partial response (PR).
Duration of Response (DOR) per RECIST V1.1 and iRECIST | Up to 5 years
  Initial and retreatment. DOR is defined as the time from the date of the first response CR/PR (whichever is first recorded) to the date of radiographical progression/death or date of censoring.
Persistence of response after discontinuation per RECIST V1.1 and iRECIST | Up to 5 years
  Initial and retreatment. Persistence of response is defined as the time from the date of treatment discontinuation to the date of radiographical progression or date of censoring.
Disease Control Rate (DCR) per RECIST V1.1 and iRECIST | Up to 5 years
  Initial and retreatment. DCR is defined as the proportion of participants for each dose level whose best overall response is rated as confirmed CR, PR or stable disease (SD).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Global Development, Inc.
Locations (32):
- United States (20):
  - Arizona Clinical Research Cent, Tucson, Arizona
  - University of California, Sacramento, California
  - University of Florida, Davis C, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa Hospitals, Iowa City, Iowa
  - Henry Ford Health System, Detroit, Michigan
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Comprehensive Cancer Nevada, Las Vegas, Nevada
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - Icahn school of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Hollings Cancer Center, Charleston, South Carolina
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Multicare Regional Cancer Center Tacoma, Tacoma, Washington
- Canada (3):
  - Site CA15002, Montreal
  - Site CA15005, Montreal
  - Site CA15004, Ontario
- South Korea (7):
  - Site KR82002, Chungcheongbukdo
  - Site KR82005, Daegu
  - Site KR82001, Gyeonggi-do
  - Site KR82003, Seoul
  - Site KR82004, Seoul
  - Site KR82006, Seoul
  - Site KR82007, Seoul
- Taiwan (2):
  - Site TW88603, Taichung
  - Site TW88604, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/1951-CL-0101/
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14537&tenant=MT_AST_9011